CLINICAL TRIAL: NCT06745960
Title: Effect of Electrical Stimulation on Painful Forward Head and Protracted Shoulder Posture in Adolescents
Brief Title: Effect of Electrical Stimulation on Forward Head Posture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yosra mostafa mohamed ali, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: forward head posture; P.T.REC/012/005173 (Registry Identifier: research ethical committee)
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Forward Head Posture; Rounded Shoulder Posture
Keywords: electrical stimulation; interferential current; adolescence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): study group (interferential current )
  Interventions: Device: electrical muscle stimulation device (EMS gymna); Other: physical therapy program
- physical therapy exercises group (Placebo Comparator): control group (exercise group)
  Interventions: Other: physical therapy program

INTERVENTIONS:
Device: electrical muscle stimulation device (EMS gymna) — muscle stimulant device
  Arms: intervention group
Other: physical therapy program — neck exercises

SUMMARY:
The study aims are:

1. To investigate the effect of electrical stimulation (interferential current) on forward head posture and protracted shoulder in adolescents.
2. To investigate the effect of electrical stimulation on cervical pain, cervical ROM, neck muscle strength, and quality of life in adolescents with forward head posture and protracted shoulder.

DETAILED DESCRIPTION:
Forward head posture (FHP) is commonly defined as the protrusion of the head in the sagittal plane so that the head is placed anterior to the trunk. It can occur because of anterior translation of the head, and it is claimed to be associated with an increase in upper cervical extension, lower cervical flexion, or both.

Patients with FHP often experience neck pain and disability, it is associated with shortening of the upper trapezius, the posterior cervical extensor muscles, the sternocleidomastoid muscle, and levator scapulae muscle. Thus, FHP may contribute to neck and shoulder pain.

The prolonged uses of mobile phones and computers have led to a variety of musculoskeletal disorders, especially related to the neck as: Forward Head Posture (FHP), rounded shoulders (RS), upper cross syndrome, mechanical neck pain etc. FHP is one in which the upper cervical convexity is increased and the lower cervical convexity is decreased causing anterior weight bearing of the cervical spine. It is also known as Scholar's neck or Reading neck.

Electrical muscle stimulation (EMS) has been used as a complementary training method, applied either locally or to the whole body. It activates muscles artificially through various electrical current forms, which are delivered through electrodes on the target muscles.

Interferential current (IFC) is an established therapy which is used to treat pain and also effective for providing relaxation of muscles. The application of IFC at the medium frequency which suggests higher penetration of the electrical stimulation in the tissue by reducing tissue impedance

ELIGIBILITY:
Inclusion Criteria:

* Girls aged between (15-18) years old.
* Normal weight with BMI ranging from (16-25).
* Adolescents with mild and moderate forward head posture(FHP).
* Adolescents with mild and moderate neck pain.
* Adolescents with protracted shoulder.

Exclusion Criteria:

* Cervical disc.
* Previous Shoulder trauma within last 6months.
* Shoulder surgery.
* Cervical fracture.
* Congenital posture deformity.
* Inflammatory disease, spinal tumor, spinal compression, spinal cord infection.
* Taking any medication for pain

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
shoulder angle (SA) | From enrollment to the end of treatment at 8 weeks
  To measure Shoulder Angle (SA) of rounded shoulder, a line from anterolateral aspect of acromion to C7 will be taken and a horizontal line from anterolateral aspect of acromion , it will be considered as forward shoulder when the angle is 52 degree or less.
craniovertebral angle (CVA) | From enrollment to the end of treatment at 8 weeks
  To measure Craniovertebral Angle (CVA) of forward head posture, a line from C7 to tragus of the ear will be taken and a horizontal line from C7 (the normal CVA more than 50 degree).
head tilt angle (HTA) | From enrollment to the end of treatment at 8 weeks
  To measure head tilt angle (HTA) or cranial angle (CA) the angle of the line between the canthus of the eye and horizontal line from the tragus, the head tilt angles is 17.74 ± 4.9 degrees in people with normal head posture.
head position angle (HPA) | From enrollment to the end of treatment at 8 weeks
  To measure head position angle (HPA) angle between the tragus manubrium line and the line extending from the center point of chin to the tragus, the angle is 38.1 ± 4.9 degrees in people with normal head posture.

SECONDARY OUTCOMES:
Pain sensation | From enrollment to the end of treatment at 8 weeks
  pain will be measured by visual analogue scale (VAS) , it is a numeric scale where 0 means no pain and 10 mean maximum pain.
cervical range of motion | From enrollment to the end of treatment at 8 weeks
  cervical rang of motion will be measured by goniometer, where the normal angles for each movement are Flexion 60 degree , Hyperextension 75 degree, Lateral Flexion 45 degree, Rotation 80 degree.
neck muscles strength | From enrollment to the end of treatment at 8 weeks
  neck muscles strength will be measured by hand held dynamometer, strength is measured in units of force per unit area. The unit is kilogram (force) per square cm (kg/cm^2)

CONTACTS AND LOCATIONS:
Overall Officials: asmaa O SAYED, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elgendy MH, Ghaffar MAA, Sabbahi SAE, Abutaleb EES, Elsayed SEB. Efficacy of head postural correction program on craniovertebral angle, scapular position, and dominant hand grip strength in forward head posture subjects: A randomized controlled trial. Physiother Res Int. 2024 Jul;29(3):e2093. doi: 10.1002/pri.2093. PMID 38780139
- [Background] Titcomb DA, Melton BF, Miyashita T, Bland HW. Evidence-Based Corrective Exercise Intervention for Forward Head Posture in Adolescents and Young Adults Without Musculoskeletal Pathology: A Critically Appraised Topic. J Sport Rehabil. 2022 Feb 16;31(5):640-644. doi: 10.1123/jsr.2021-0381. Print 2022 Jul 1. PMID 35172275
- See also: effect of electrical muscle stimulation — https://www.medicalnewstoday.com/articles/electrical-muscle-stimulation
- See also: image of angles needed to be measured in this study — https://images.app.goo.gl/TZyc6FqfEX1GASDm8